CLINICAL TRIAL: NCT07207915
Title: Analysis of Integrated Clinical, Laboratory and Prognostic Data of Neonates With Necrotizing Enterocolitis
Acronym: ACLPNEC
Status: Completed | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hu Hao, Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: EK-NEC20250701; 2025A1515012514 (Other Grant/Funding Number: Natural Science Foundation of Guangdong Province)
Record Dates: First submitted 2025-09-21; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Necrotizing Enterocolitis
Keywords: necrotizing enterocolitis; Lactate; Intestinal perforation; Mortality; nSOFA
MeSH Terms: conditions — Enterocolitis, Necrotizing; Intestinal Perforation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- Mild NEC group: Bell's stage I and IIa
  Interventions: Other: Observational retrospective cohort study
- Severe NEC group: Bell's stage IIb and III
  Interventions: Other: Observational retrospective cohort study
- NIP group: non-intestinal perforation in surgical NEC
  Interventions: Other: Observational retrospective cohort study
- PNEC group: Perforated necrotizing enterocolitis
  Interventions: Other: Observational retrospective cohort study

INTERVENTIONS:
Other: Observational retrospective cohort study — Observational retrospective cohort study, data collection was performed via structured extraction from electronic medical records: Includingclinical characteristics, metabolic indicators, laboratory parameters, prognosis, and outcomes.

SUMMARY:
This is a retrospective study led by The Sixth Affiliated Hospital, Sun Yat-sen University, focusing on newborns diagnosed with necrotizing enterocolitis (NEC)-a serious gastrointestinal disease that threatens newborns' lives-between January 2023 and June 2025.

Purpose of the study: NEC can lead to severe conditions like bowel perforation or even death, and it's hard for doctors to spot high-risk babies early with current tools. This study aims to analyze the babies' clinical information (e.g., birth weight, symptoms like belly swelling or bloody stools), blood test results (e.g., lactate levels, white blood cell counts), and organ function scores (nSOFA scores) to find indicators that can predict whether NEC will get worse or cause death.

Questions the study tries to answer: Can combining metabolic indicators (like lactate), blood test parameters, and organ function scores better predict if a newborn with NEC will develop perforated NEC (a more severe form where the bowel has holes) or die during hospitalization? Are these combined indicators more reliable than single indicators alone? Study hypothesis: We guess that integrating metabolic markers (such as lactate), blood routine parameters, and nSOFA scores will be more accurate than using any single indicator to predict the progression of NEC and the risk of death in affected newborns.

DETAILED DESCRIPTION:
1. Study Rationale Necrotizing Enterocolitis (NEC) is a life-threatening gastrointestinal disorder primarily affecting very low birth weight (VLBW) neonates (incidence: 5-12%). Around 20-40% of cases progress to severe disease requiring surgery, and survivors often face long-term complications (e.g., short-bowel syndrome, neurodevelopmental impairments). Despite advances in neonatal care, early identification of high-risk patients remains challenging due to nonspecific clinical/radiographic signs and insufficiently sensitive/specific conventional biomarkers.

   NEC pathophysiology involves intestinal ischemia-reperfusion injury, excessive immune activation, and microbial dysbiosis. Serum lactate (a marker of hypoperfusion/anaerobic metabolism) correlates with NEC severity but lacks specificity; peripheral blood cell (CBC) indices are accessible but understudied in combination with lactate. The Neonatal Sequential Organ Failure Assessment (nSOFA) score predicts overall NEC mortality but fails to stratify risk for perforated NEC (PNEC), a high-risk subtype. This study aims to address gaps by integrating metabolic (lactate), hematologic (CBC), and organ dysfunction (nSOFA) metrics for NEC prognosis.
2. Study Design and Conduct This is a retrospective cohort study conducted at the Sixth Affiliated Hospital, Sun Yat-sen University, approved by the institutional ethics committee and compliant with the Helsinki Declaration. The study period is January 1, 2023-June 30, 2025; eligible participants are identified via retrospective review of electronic medical records (EMRs), with data extracted in a structured manner.
3. Data Collection

   Structured EMR extraction captures key variables:

   Neonatal history: Sex, gestational age, birth weight, birth asphyxia (Apgar scores), small for gestational age (SGA) status, preterm complications (e.g., patent ductus arteriosus [PDA], respiratory distress syndrome [RDS]), feeding pattern, mechanical ventilation use.

   Maternal history: Delivery mode, chorioamnionitis, premature rupture of membranes.

   NEC-related parameters: Bell's staging, clinical manifestations (e.g., abdominal distension, pneumoperitoneum), complications (sepsis, shock), therapeutic interventions (surgery), in-hospital mortality.

   Laboratory/organ dysfunction indicators: Serum lactate (at NEC onset), CBC parameters (WBC, neutrophils, lymphocytes, platelets) and derived inflammatory indices, nSOFA score (at NEC onset).
4. Statistical Analysis

   Analyses use SPSS 26.0 and GraphPad Prism 9.0:

   Data expression: Normally distributed variables (mean ± SD), skewed variables (median [IQR]), categorical variables (frequency %).

   Intergroup comparisons: Chi-square/Fisher's exact test (categorical), t-test/Mann-Whitney U test (continuous).

   Multivariate logistic regression: Includes variables with p<0.05 from univariate analysis to identify independent predictors.

   Mediation analysis (PROCESS macro 4.1, 1000 bootstraps): Decomposes total effects into direct/indirect paths.

   ROC curve analysis: Evaluates predictive performance of single/combined biomarkers (AUC as metric). All tests are two-tailed; p<0.05 is significant.
5. Study Objectives Primary: Identify indicators predicting NEC progression (PNEC) and in-hospital mortality via analysis of clinical, metabolic, and laboratory data.

   Secondary: Explore integrated biomarkers for NEC severity stratification (e.g., Bell's staging, surgical need) to optimize clinical decision-making.
6. Participant Protection All data are de-identified before analysis and stored in a password-protected database (accessible only to the study team). Informed consent is obtained from participants' legal representatives, who are informed of the right to withdraw at any time without penalty.

ELIGIBILITY:
Inclusion Criteria:

* (1) Diagnosis of NEC and having undergone surgical treatment, confirmed by clinical manifestations (e.g., abdominal distension, bloody stools), radiological evidence (pneumatosis intestinalis, portal venous gas, or pneumoperitoneum), and pathological examination in accordance with established guidelines; (2) Availability of complete medical records for data extraction.

Exclusion Criteria:

* (1) Congenital gastrointestinal malformations (e.g., intestinal atresia, Hirschsprung's disease) or spontaneous intestinal perforation; (2) Hereditary metabolic disorders; (3) Incomplete clinical data or refusal of participation.

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: In this study, a retrospective analysis was conducted on 400 enrolled neonates with necrotizing enterocolitis (NEC), with data collected at The Sixth Affiliated Hospital, Sun Yat-sen University from January 2023 to June 2025.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
Occurrence of perforated necrotizing enterocolitis | Day 1 up to 3 months
  Occurrence of perforated necrotizing enterocolitis
In-hospital mortality | Day 1 up to 3 months
  In-hospital mortality

SECONDARY OUTCOMES:
Bell's Staging System for Necrotizing Enterocolitis (NEC) | Day 1 up to 3 months
  The Bell staging system is a standardized clinically validated classification tool for assessing the severity of necrotizing enterocolitis (NEC), integrating clinical manifestations, imaging, and laboratory data. Assessment criteria include: clinical symptoms (e.g., abdominal distension, bloody stools, feeding intolerance, shock); imaging findings (abdominal X-ray showing intestinal pneumatosis, portal venous gas, pneumoperitoneum, etc.); and laboratory results (thrombocytopenia, metabolic acidosis, etc.). Staging is determined by the research team through review of neonates' complete clinical, imaging, and laboratory records (extracted per the study's structured protocol) to ensure alignment with established Bell staging criteria.
Incidence of Surgical Necrotizing Enterocolitis (NEC) | Day 1 up to 3 months
  "Surgical NEC" in this study refers to necrotizing enterocolitis (NEC) cases requiring surgical intervention. Its assessment relies on abdominal X-ray, abdominal ultrasound, and Bell's Staging System (as referenced in the Study Protocol with Statistical Analysis Plan.docx), with data extracted from neonates' electronic medical records per the protocol's data collection framework.
  Eligibility for classifying a case as surgical NEC is determined by: 1) Abdominal X-ray/ultrasound findings indicating severe NEC progression (e.g., pneumoperitoneum, unresponsive extensive pneumatosis intestinalis); 2) Bell's Staging (assessed per study criteria) confirming Stage III (Advanced NEC) - both consistent with clinical standards for initiating NEC-related surgery. The study team reviews these imaging results and staging data to confirm surgical NEC uniformly.

CONTACTS AND LOCATIONS:
Overall Officials: Hu Hao, Doctor, Study Chair — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospial, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lewis AN, de la Cruz D, Wynn JL, Frazer LC, Yakah W, Martin CR, Yang H, Itriago E, Unger J, Hair AB, Miele J, Sullivan BA, Husain A, Good M. Evaluation of the Neonatal Sequential Organ Failure Assessment and Mortality Risk in Preterm Infants with Necrotizing Enterocolitis. Neonatology. 2022;119(3):334-344. doi: 10.1159/000522560. Epub 2022 Mar 21. PMID 35313308
- [Result] Li B, Chen Y, Yang Z, Sun X, Tian C, Liu J, Yuan L, Dai K. Lactate/albumin ratio as a prognostic biomarker for in-hospital mortality in pediatric patients with necrotizing enterocolitis. BMC Pediatr. 2025 Feb 4;25(1):93. doi: 10.1186/s12887-025-05439-5. PMID 39905329
- [Result] El-Abd Ahmed A, Hassan MH, Abo-Halawa N, Abdel-Razik GM, Moubarak FA, Sakhr HM. Lactate and intestinal fatty acid binding protein as essential biomarkers in neonates with necrotizing enterocolitis: ultrasonographic and surgical considerations. Pediatr Neonatol. 2020 Oct;61(5):481-489. doi: 10.1016/j.pedneo.2020.03.015. Epub 2020 Apr 5. PMID 32336643
- [Result] Kislal FM, Polat CC, Ergul E, Acikalin AA, Guven D, Gundogan E, Sarici D. Can lactate be valuable in early diagnosis and prognosis of neonatal sepsis? Niger J Clin Pract. 2023 Sep;26(9):1319-1325. doi: 10.4103/njcp.njcp_54_23. PMID 37794545
- [Result] Wang Y, Lai L, Zhang Q, Zheng L. Lactate acid level and prognosis of neonatal necrotizing enterocolitis: a retrospective cohort study based on pediatric-specific critical care database. J Pediatr (Rio J). 2023 May-Jun;99(3):278-283. doi: 10.1016/j.jped.2022.11.005. Epub 2022 Dec 16. PMID 36535423
- [Result] Roberts AG, Younge N, Greenberg RG. Neonatal Necrotizing Enterocolitis: An Update on Pathophysiology, Treatment, and Prevention. Paediatr Drugs. 2024 May;26(3):259-275. doi: 10.1007/s40272-024-00626-w. Epub 2024 Apr 2. PMID 38564081
- [Result] Kim JH, Sampath V, Canvasser J. Challenges in diagnosing necrotizing enterocolitis. Pediatr Res. 2020 Aug;88(Suppl 1):16-20. doi: 10.1038/s41390-020-1090-4. PMID 32855507
- [Result] Clyman RI, Jin C, Hills NK. A role for neonatal bacteremia in deaths due to intestinal perforation: spontaneous intestinal perforation compared with perforated necrotizing enterocolitis. J Perinatol. 2020 Nov;40(11):1662-1670. doi: 10.1038/s41372-020-0691-4. Epub 2020 May 20. PMID 32433511
- [Result] Fitzgibbons SC, Ching Y, Yu D, Carpenter J, Kenny M, Weldon C, Lillehei C, Valim C, Horbar JD, Jaksic T. Mortality of necrotizing enterocolitis expressed by birth weight categories. J Pediatr Surg. 2009 Jun;44(6):1072-5; discussion 1075-6. doi: 10.1016/j.jpedsurg.2009.02.013. PMID 19524719
- [Result] Sakellaris G, Partalis N, Dede O, Alegakis A, Seremeti C, Korakaki E, Giannakopoulou C. Gastrointestinal perforations in neonatal period: experience over 10 years. Pediatr Emerg Care. 2012 Sep;28(9):886-8. doi: 10.1097/PEC.0b013e31826beb0c. PMID 22929145
- [Result] Chen M, Feng W, Hou J, Die X, Guo Z, Wang Y. Effect of gestational age on clinical features in necrotizing enterocolitis-associated intestinal perforation. Front Pediatr. 2025 Jan 6;12:1452207. doi: 10.3389/fped.2024.1452207. eCollection 2024. PMID 39834496
- [Result] Imren C, Vlug LE, de Koning BAE, Diertens T, Snel HE, Suurland J, Swarte RMC, Vermeulen MJ, Keyzer-Dekker CMG. Necrotizing Enterocolitis in a Dutch Cohort of Very Preterm Infants: Prevalence, Mortality, and Long-Term Outcomes. Eur J Pediatr Surg. 2022 Feb;32(1):111-119. doi: 10.1055/s-0041-1741544. Epub 2022 Jan 10. PMID 35008115
- [Result] Butler V, Treluyer L, Patkai J, Biset A, Jarreau PH, Ancel PY, Roze JC, Marchand-Martin L, Durox M, Lapillonne A, Picaud JC, Mitanchez D, Tscherning C, Biran V, Cambonie G, Lopez E, Hascoet JM, Desfrere L, Chollat C, Zana-Taieb E, Torchin H. Mortality and neurodevelopmental outcomes at 2 years' corrected age of very preterm infants with necrotising enterocolitis or spontaneous intestinal perforation: The EPIPAGE-2 cohort study. Eur J Pediatr. 2024 Sep;183(9):4019-4028. doi: 10.1007/s00431-024-05675-4. Epub 2024 Jul 2. PMID 38955846
- [Result] Vaidya R, Yi JX, O'Shea TM, Jensen ET, Joseph RM, Shenberger J, Gogcu S, Wagner K, Msall ME, Thompson AL, Frazier JA, Fry R, Singh R; ELGAN-ECHO Study Investigators. Long-Term Outcome of Necrotizing Enterocolitis and Spontaneous Intestinal Perforation. Pediatrics. 2022 Nov 1;150(5):e2022056445. doi: 10.1542/peds.2022-056445. PMID 36200375
- [Result] Bazacliu C, Neu J. Necrotizing Enterocolitis: Long Term Complications. Curr Pediatr Rev. 2019;15(2):115-124. doi: 10.2174/1573396315666190312093119. PMID 30864508
- [Result] Jiang S, Yan W, Li S, Zhang L, Zhang Y, Shah PS, Shah V, Lee SK, Yang Y, Cao Y. Mortality and Morbidity in Infants <34 Weeks' Gestation in 25 NICUs in China: A Prospective Cohort Study. Front Pediatr. 2020 Feb 13;8:33. doi: 10.3389/fped.2020.00033. eCollection 2020. PMID 32117838

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT07207915/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT07207915/ICF_001.pdf